CLINICAL TRIAL: NCT02571985
Title: Clinical Study to Evaluate the Safety and Effectiveness of the Zenith® Branch Endovascular Graft-Iliac Bifurcation With the ConnectSX™
Brief Title: PRESERVE-Zenith® Iliac Branch System Clinical Extended Study
Status: No longer available | Type: Expanded Access
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-625 CA-P1
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Aorto-iliac Aneurysms; Iliac Aneurysms
Keywords: Zenith aortoiliac aneurysm; iliac aneurysm; branch; connections; endovascular graft; graft-iliac bifurcation; Aneurysm; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Iliac Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases

INTERVENTIONS:
Device: Zenith® Branch Endovascular Graft-Iliac Bifurcation System — Zenith® Branch Endovascular Graft-Iliac Bifurcation (Branch Graft) with the ConnectSX™
  Other Names: Endovascular repair for aortoiliac or iliac aneurysm

SUMMARY:
The PRESERVE-Zenith® Iliac Branch System Clinical Study is a clinical trial to collect confirmatory safety and effectiveness data on the Zenith® Branch Endovascular Graft-Iliac Bifurcation System. This system is made up of two devices: the Zenith® Branch Endovascular Graft-Iliac Bifurcation and the ConnectSX™ covered stent in the treatment of aorto-iliac and iliac aneurysms

ELIGIBILITY:
Inclusion Criteria:

* An aortioiliac or iliac aneurysm
* An unsuitable distal sealing site for a traditional Zenith iliac leg graft within the common lilac artery

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2017-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: W. Anthony Lee, MD FACS, Principal Investigator — Christine E. Lynn Heart and Vascular Institute
Locations (19):
- United States (19):
  - VA Palo Alto HCS, Palo Alto, California
  - Stanford University Medical School, Stanford, California
  - Christine E. Lynn Heart and Vascular Institute, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Massachusetts, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital East Communities, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin